CLINICAL TRIAL: NCT03311672
Title: T-Cell PET Imaging With [18F]F-AraG and Radiomics to Guide Combined Radiation and Systemic Immune Modulating Therapies
Brief Title: T-Cell PET Imaging With [18F]F-AraG in Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: University of California, San Francisco (Other)
Collaborators: CellSight Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 176513; NCI-2018-02158 (Other: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2017-10-11; First posted 2017-10-17 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 - Immunotherapy Alone (Experimental): Approximately 10 patients will be enrolled in the immunotherapy alone cohort under a larger two-year industry-funded, investigator-initiated single-institution, phase II, open-label clinical trial (NCT03217071; Pembrolizumab With and Without Radiotherapy for Non-Small Cell Lung Cancer) in which patients with stage I-IIIA non-small cell lung cancer (NSCLC) are randomized to receive two cycles of systemic immunotherapy (pembrolizumab, a PD-1 inhibitor) with or without immune-priming stereotactic radiation therapy (SRT, 12 Gy) to the lateral half of the primary lung tumor prior to resection.
  Interventions: Drug: [18F]F-Ara-G; Drug: Pembrolizumab; Radiation: PET/CT scan
- Cohort 2 - Immunotherapy with Stereotactic Radiation (Experimental): Approximately 10 patients will be enrolled in the immunotherapy with stereotactic radiation therapy cohort under a larger two-year industry-funded, investigator-initiated single-institution, phase II, open-label clinical trial (NCT03217071; Pembrolizumab With and Without Radiotherapy for Non-Small Cell Lung Cancer) in which patients with stage I-IIIA non-small cell lung cancer (NSCLC) are randomized to receive two cycles of systemic immunotherapy (pembrolizumab, a PD-1 inhibitor) with or without immune-priming stereotactic radiation therapy (SRT, 12 Gy) to the lateral half of the primary lung tumor prior to resection.
  Interventions: Drug: [18F]F-Ara-G; Drug: Pembrolizumab; Radiation: PET/CT scan

INTERVENTIONS:
Drug: [18F]F-Ara-G — Administered after two cycles of immunotherapy +/- stereotactic radiation therapy as part of the PET/CT scan.
  Other Names: 2'-deoxy-2'-[18F]fluoro-9-β-Darabinofuranosylguanine
Drug: Pembrolizumab — All study participants will receive pembrolizumab every 3 weeks, for 2 cycles.
  Other Names: Keytruda
Radiation: PET/CT scan — Scan will be done after two cycles of immunotherapy +/- stereotactic radiation therapy.

SUMMARY:
This is a single-center cross-sectional imaging study in patients with localized lung cancer undergoing immunotherapy with or without stereotactic radiation therapy as part of the companion clinical trial (NCT03217071; Pembrolizumab With and Without Radiotherapy for Non-Small Cell Lung Cancer). Each patient will undergo a single [18F]F-AraG PET exam as part of this study. [18F]F-AraG will be administered at a single time point intravenously prior to PET imaging. Whole-body PET will be acquired along with a whole body low dose CT (PET/CT) used for attenuation correction and anatomic localization of [18F]F-AraG uptake, SUV calculation, and volumetric selection for radiomic analyses.

DETAILED DESCRIPTION:
This is a single-center cross-sectional imaging study in patients with localized lung cancer undergoing immunotherapy with or without stereotactic radiation therapy as part of the companion clinical trial (NCT03217071; Pembrolizumab With and Without Radiotherapy for Non-Small Cell Lung Cancer). Each patient will undergo a single [18F]F-AraG PET exam as part of this study. [18F]F-AraG will be administered at a single time point intravenously prior to PET imaging. Whole-body PET will be acquired along with a whole body low dose CT (PET/CT) used for attenuation correction and anatomic localization of [18F]F-AraG uptake, SUV calculation, and volumetric selection for radiomic analyses.

A total of 20 patients will be enrolled over an accrual period of approximately 12 months. Approximately 10 patients will be enrolled in the immunotherapy alone cohort and approximately 10 patients will be enrolled in the immunotherapy and stereotactic radiation therapy cohort.

Patients will be evaluated one day and one week via telephone after each radiopharmaceutical injection for safety follow-up. All adverse events will be recorded. Due to the noninvasive and non-therapeutic nature of the study, potential risks of the study are anticipated to be low.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years
2. Histologically or cytologically documented stage I-IIIA non-small cell lung cancer (NSCLC)
3. Eligible for with plan to undergo immunotherapy alone or both immunotherapy and stereotactic radiation therapy as part of NCT03217071
4. In female patients, negative pregnancy test with no plans to become pregnant during the duration of the study
5. Able to provide informed consent and follow the study guidelines

Exclusion Criteria:

1. Female patients who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-26 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
The correlation between number of infiltrating CD3+ T cells/μm2 in the non-small cell lunger cancer thoracotomy specimen as quantified by immunohistochemistry and the activated T-cell concentration as determined by [18F]F-AraG PET (SUVmax) | Baseline (after two cycles of pembrolizumab)
  The correlation between number of infiltrating CD3+ T cells/μm2 in the non-small cell lunger cancer thoracotomy specimen as quantified by immunohistochemistry and the activated T-cell concentration as determined by [18F]F-AraG PET (SUVmax)

SECONDARY OUTCOMES:
The detection of out-of-target radiation-mediated immune modulation in lymph nodes using [18F]F-AraG PET | Baseline (after two cycles of pembrolizumab)
  The detection of out-of-target radiation-mediated immune modulation in lymph nodes using [18F]F-AraG PET

CONTACTS AND LOCATIONS:
Overall Officials: Sue Yom, MD, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No